CLINICAL TRIAL: NCT01672515
Title: Phase 2 Study of Remote Limb Ischemic Preconditioning on Acute Cerebral Infarction
Brief Title: Protective Effects of Remote Limb Ischemic Preconditioning on Acute Cerebral Infarction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming, Professor of Neurosurgery, Vice-President of Xuan Wu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-RIPC-cerebral infarction
Record Dates: First submitted 2012-08-19; First posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC group (Experimental): RIPC treatment was performed by the inflating tourniquets to 200mmHg on bilateral arms with 5 cycles of 5min inflation and 5min relax alternation for the total of 30 consecutive days.
  Interventions: Device: RIPC group
- Control group (Sham Comparator): RIPC sham was performed by the inflating tourniquets to 60mmHg on bilateral arms with 5 cycles of 5min inflation and 5min relax alternation for the total of 30 consecutive days.
  Interventions: Device: Control group

INTERVENTIONS:
Device: RIPC group
  Other Names: Brand name: Doctormate; Type: IPC-906X; Productor: Beijing Renqiao Institute of Neuroscience
  Arms: RIPC group
Device: Control group
  Other Names: Brand name: Doctormate; Type: modified version of IPC-906X; Productor: Beijing Renqiao Institute of Neuroscience
  Arms: Control group

SUMMARY:
Stroke is one of the three leading causes of human death, and a major cause of adult disability. Our pre-clinical studies confirmed that ischemic preconditioning can prevent cerebral infarction. Animal studies confirmed that ischemic postconditioning can reduce infarct size of cerebral infarction. Investigators hypothesized that postconditioning would reduce infarct volume of ischemic stroke patients.

DETAILED DESCRIPTION:
This study explored the neuroprotective effects of post-positioning on ischemic stroke patients with randomized, double-blinded and controlled method. Patients are divided into experimental and placebo groups to receive remote ischemic post-conditioning for 30 days. Remote ischemic post-conditioning is performed by the inflating tourniquets to certain extents on bilateral arms with 5 cycles of 5min inflation and 5min relax alternation for the total of 30 consecutive days. It is 200mmHg for RIPC group and 60mmHg for control group. Evaluation parameters include CRP, TNF-α, ICAM-1 and GFAP in blood at 0, 3, 7, 15 and 30 days after treatment; and MRI at 0 and 30 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age between 40 to 80 Years
2. Ischemic cerebrovascular disease within 6 hours
3. National Institutes of Health Stroke Scale(NIHSS) score 0-15,and Modified Rankin Scale(mRS) score 0-4
4. Cranial CT to rule out the the cerebral hemorrhage
5. Written informed consent was

Exclusion Criteria:

1. Cerebral hemorrhage
2. Other parts of the active bleeding disease
3. Atrial fibrillation
4. Moyamoya disease or vasculitis
5. Hereditary disease, such as with CADASIL, FABRY, mitochondrial myopathy
6. Out coagulation disorder
7. Severe lesions of severe liver and kidney disease, malignancy or other systemic
8. Cannot tolerate BLIPC or without informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Local tissue damage 30 days after RIPC treatment | 30 days after RIPC treatment
  Evaluated by the doctor blinded to the study protocol, including: local edema, redness, skin breakage
Levels of plasma biomarkers assay right before RIPC treatment | right before RIPC treatment (within 24hrs)
  levels of CRP、TINF-α、slCAM-1 and GFAP
Levels of plasma biomarkers assay 3 days after RIPC treatment. | 3 days after RIPC treatment.
  levels of CRP、TINF-α、slCAM-1 and GFAP
Levels of plasma biomarkers assay 15 days after RIPC treatment. | 15 days after RIPC treatment.
  levels of CRP、TINF-α、slCAM-1 and GFAP
Levels of plasma biomarkers assay 30 days after RIPC treatment | 30 days after RIPC treatment
  levels of CRP、TINF-α、slCAM-1 and GFAP
Levels of plasma biomarkers assay right after RIPC treatment | right after RIPC treatment (within 24hrs)
  levels of CRP、TINF-α、slCAM-1 and GFAP

SECONDARY OUTCOMES:
Infarct volume evaluation before RIPC treatment. | Acute phase of ischemic stroke, and before RIPC treatment
  MRI evaluation of infarct volume in ischemic stroke patients before RIPC treatment.
Infarct volume after RIPC treatment in ischemic stroke patients | 30 days after RIPC treatment in ischemic stroke patients
  Infarct volume evaluation in ischemic stroke patients after 30 RIPC treatment